CLINICAL TRIAL: NCT06278909
Title: Trigeminal Nerve Stimulation in Treatment-resistant Generalized Anxiety Disorder: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Rafael Freire (Other)
Responsible Party: Sponsor-Investigator, Dr. Rafael Freire, Associate Professor, Department of Psychiatry, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6036699
Record Dates: First submitted 2024-02-09; First posted 2024-02-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: This is a traditional feasibility study, which evaluates preliminary safety and effectiveness information. It does not meet the definition of a "device feasibility" study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active stimulation (Experimental): Trigeminal nerve stimulation will occur by placement of electrodes (1.25" silver electrodes Bio-Flex BF4, Biotens/Vermed, Buffalo, New York, USA) bilaterally on the V1 branches of the trigeminal nerve (CNV) located on the forehead. Current will be generated from the EMS 7500 stimulator (TENS Products, Inc., Granby, CO) (Class II medical device) and will be set to a level that is clearly perceptible by each patient (i.e. tingling sensation) but not uncomfortable or painful. Current level will be determined for each patient at baseline and will likely be between 4-6 milliampere (mA). Active stimulation will occur at 120 Hz with a 250 μs pulse width and with a duty cycle of 30 seconds on to 30 seconds off.
  Interventions: Device: Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation — Active trigeminal nerve stimulation

SUMMARY:
This is a feasibility study for trigeminal nerve stimulation (TNS) in patients with treatment-resistant generalized anxiety disorder (TR-GAD). Ten participants will receive TNS for 8 weeks as an augmentation strategy to pharmacological treatment for generalized anxiety disorder (GAD).

* The primary objective is to ascertain if TNS is a safe and well-tolerated treatment for patients with TR-GAD.
* The secondary objective will be to monitor changes in GAD symptom severity throughout the study.

Results from this study will inform a randomized controlled trial to be conducted in the future.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5) criteria for generalized anxiety disorder.
* Subjects on a stable dose of an selective serotonin reuptake inhibitor (SSRI) or serotonin and noradrenaline reuptake inhibitor (SNRI) for at least 8 weeks.
* Treatment-resistant - treatment resistance will be defined as lack of response to at least two drugs, from two different classes of drugs considered first-line or second-line for GAD. Only trials lasting at least 8 weeks, and with at least the minimum effective dose of the given medication will be considered failed trials.

Exclusion Criteria:

* Moderate to severe major depressive disorder
* Moderate to high suicidality
* Diagnosis of obsessive compulsive disorder (OCD), PTSD, bipolar disorder, schizophrenia, schizoaffective disorder, personality disorders, substance use disorders, intellectual disabilities and dementia or other neurological diseases including trigeminal neuralgia
* Pregnant or breastfeeding women
* Participants who are experiencing seizures
* Implanted vagal nerve stimulation (VNS) or other electrical devices
* Participants who are already undergoing transcutaneous electrical nerve stimulation
* Consumption of cannabis, any cannabis by-products, illicit drugs, or alcohol above 3 drinks per week
* Consumption of natural health products that may affect anxiety or depression symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Throughout the study, 8 weeks
  Monitor participants for treatment-emergent adverse events and serious adverse events.
Incidence of treatment-emergent side effects measured with the NSEC | Baseline visit, 4-week visit and 8-week visit.
  Monitor participants for minor treatment-emergent side effects measured with the Neurostimulation Side-Effect Checklist (NSEC).
  NSEC is a list of 31 possible side effects from neurostimulation or from antidepressants. Each item is rated from 0 (absent) to 3 (severe).
Response to treatment defined by CGI-I score below 3 | 4-week visit and 8-week visit.
  Response to treatment, which will be defined as a score of 1 or 2 on the Clinical Global Impression - Improvement (CGI-I) scale.
  CGI-I is a clinician administered one-item clinical scale rated from 1 (very much improved) to 7 (very much worse). Not assessed would confer score 0.

SECONDARY OUTCOMES:
Remission defined by CGI-S score below 3 | 4-week visit and 8-week visit.
  Remission will be defined as a score of 1 or 2 on the Clinical Global Impression - Severity (CGI-S) scale.
  CGI-S is a clinician administered one-item clinical scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Not assessed would confer score 0.
Change in anxiety severity measured by CGI-S | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for CGI-S by comparing the scores in each visit. CGI-S is a clinician administered one-item clinical scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Not assessed would confer score 0.
Change of anxiety symptoms measured with GAD-7 | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for Generalized Anxiety Disorder 7-item scale (GAD-7) by comparing the scores in each visit.
  GAD-7 is a self-rated 7-item scale, each item is rated from 0 (not at all) to 3 (nearly every day).
Change of anxiety symptoms measured with PSWQ | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for Penn State Worry Questionnaire (PSWQ) by comparing the scores in each visit.
  PSWQ is a self-rated 16-item scale, each item is rated from 1 (not at all typical of me) to 5 (very typical of me).
Change of anxiety symptoms measured with BAI | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for Beck Anxiety Inventory (BAI) by comparing the scores in each visit.
  BAI is a self-rated 21-item scale, each item is rated from 0 (not at all) to 3 (severely - it bothered me a lot).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Freire, MD PhD, Principal Investigator — Department of Psychiatry, Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook IA, Abrams M, Leuchter AF. Trigeminal Nerve Stimulation for Comorbid Posttraumatic Stress Disorder and Major Depressive Disorder. Neuromodulation. 2016 Apr;19(3):299-305. doi: 10.1111/ner.12399. Epub 2016 Jan 28. PMID 26818103
- [Background] Cook IA, Schrader LM, Degiorgio CM, Miller PR, Maremont ER, Leuchter AF. Trigeminal nerve stimulation in major depressive disorder: acute outcomes in an open pilot study. Epilepsy Behav. 2013 Aug;28(2):221-6. doi: 10.1016/j.yebeh.2013.05.008. Epub 2013 Jun 14. PMID 23773978
- [Background] Freire RC, Cabrera-Abreu C, Milev R. Neurostimulation in Anxiety Disorders, Post-traumatic Stress Disorder, and Obsessive-Compulsive Disorder. Adv Exp Med Biol. 2020;1191:331-346. doi: 10.1007/978-981-32-9705-0_18. PMID 32002936
- [Background] Trevizol AP, Shiozawa P, Sato IA, Calfat EL, Alberto RL, Cook IA, Medeiros HH, Cordeiro Q. Trigeminal Nerve Stimulation (TNS) for Generalized Anxiety Disorder: A Case Study. Brain Stimul. 2015 May-Jun;8(3):659-60. doi: 10.1016/j.brs.2014.12.009. Epub 2014 Dec 31. No abstract available. PMID 25650095